CLINICAL TRIAL: NCT01588002
Title: A Study to Evaluate the Potential Drug-Drug Interaction Between Efavirenz and Danoprevir With Low Dose Ritonavir When Administered Together in Healthy Adult Volunteers
Brief Title: A Study of Potential Drug-Drug Interaction Between Efavirenz and Danoprevir With Low Dose Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28103
Record Dates: First submitted 2012-04-19; First posted 2012-04-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; efavirenz; Ritonavir

ARMS (3):
- A danoprevir+ritonavir (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir
- B efavirenz (Active Comparator)
  Interventions: Drug: efavirenz
- C combination (Experimental)
  Interventions: Drug: danoprevir; Drug: efavirenz; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — multiple oral doses
  Arms: A danoprevir+ritonavir; C combination
Drug: efavirenz — multiple oral doses
  Arms: B efavirenz; C combination
Drug: ritonavir — multiple oral doses
  Arms: A danoprevir+ritonavir; C combination

SUMMARY:
This phase 1, randomized, open-label, multiple-dose, 2-sequence, 2-period crossover study will evaluate potential drug-drug interaction between efavirenz and danoprevir with low-dose ritonavir in healthy volunteers. In Period 1. subjects will be randomized to receive multiple oral doses of either danoprevir with ritonavir or efavirenz for 14 days. In Period 2, all subjects will receive multiple oral doses of the combination danoprevir with ritonavir and efavirenz for 14 days. Anticipated time on study treatment is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female non-smoking subjects, 18 to 55 years of age
* Healthy status will be defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Medical history without major, recent or ongoing pathology
* Weight >/= 50.0 kg
* Body mass index (BMI) 18.0 - 32.0 kg/m2

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* History of any clinically significant medical condition which may impact the safety of the participant
* Positive results for drugs of abuse at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection
* Current smokers or subjects who have discontinued smoking less than 6 months prior to first dose of study medication
* Use of hormonal contraceptives (e.g. birth control pill, patches, or injectable, implantable devices) within 30 days before the first dose of study medication
* Use of investigational drug or device within 30 days of the first dose of study medication (6 months for biologic therapies) or 5 half-lives of the investigational drug, whichever is longer
* History of drug-related allergic reaction
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average; alcohol consumption will be prohibited 72 hours prior to entry in the clinical site center and throughout the entire study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of efavirenz, danoprevir and ritonavir in coadministration: Cmax | Pre-dose and up to 24 hours post-dose on Days 14 and 28
Pharmacokinetics of efavirenz, danoprevir and ritonavir in coadministration: Area under the concentration-time curve (AUC) | Pre-dose and up to 24 hours post-dose on Days 14 and 28

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States